CLINICAL TRIAL: NCT01845051
Title: Is There a Comorbidity Between Migraine and Allergic Rhinitis?
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Işıl Adadan Güvenç, MD, ENT Specialist, Baskent University
Other Study IDs: CC-01
Record Dates: First submitted 2013-04-29; First posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Migraine; Allergic Rhinitis
Keywords: Migraine; allergic rhinitis; Specific Immunoglobulin E (IgE); nasal symptoms; signs of allergy.
MeSH Terms: conditions — Migraine Disorders; Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Migraine group: Patients diagnosed with migraine
- Healthy group: Healthy subjects with no migraine as control

SUMMARY:
The researchers investigated the relationship between migraine and allergy. For this purpose, the researchers designed a controlled study to evaluate nasal symptoms and signs; and to perform Specific Immunoglobulin E (IgE) measurements in migraine patients and healthy subjects. According to these results the prevalence of allergic rhinitis in migraine group was planned to be compared to that of the healthy controls, statistically.

ELIGIBILITY:
Inclusion Criteria:

* patients with migraine

Exclusion Criteria:

* other neurologic disorders that may contribute to headaches, such as stroke, cerebral palsy, trigeminal neuralgia, and seizure disorder
* also acute and chronic sinusitis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Migraine patients attending neurology clinic and healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Specific Immunoglobulin E (IgE) | 1 day
  Blood samples were taken from study and control group for the determination of Specific IgE panel against six different allergens: (1) fungi, (2) grass pollens, (3) tree pollens, (4) wild herbs, (5) mite 1, (6) mite 2. For all of specific IgE panels, <0,7 RU/ml was negative; and >0,7 RU/ml was Positive.
Nasal Symptom Scores | 1 day
  Symptoms were assessed with a questionnaire for the presence and severity of allergic rhinitis (AR) symptoms on a scale of 0-3 (0 = none, 1 = mild, 2 = moderate, 3 = severe). Symptoms of AR (Nasal discharge, nasal congestion, itching and sneezing) were graded between 0-3.

OTHER OUTCOMES:
İnferior turbinate color and edema | 1 day
  inferior concha colour (0=natural, 1=pale, 2=bluish and 3=severely pale or bluish) and turbinate edema were assessed during ENT examination on 0-3 scale (0 = no, 1 = mild, 2 = moderate, 3 = severe).